CLINICAL TRIAL: NCT06102031
Title: A Multicenter, Randomized, Controlled Clinical Study to Evaluate the Effectiveness of Using the Noninvasive Lung Fluid Monitoring System Based on Remote Dielectric Sensing in Guiding the Treatment of Heart Failure
Brief Title: Clinical Study on the Noninvasive Lung Fluid Monitoring System in Guiding the Treatment of Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V2.0
Record Dates: First submitted 2023-10-11; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized Arm-Treatment Group (Experimental): Management of subjects based on lung fluid content derived from the ReDS™ system.
  All subjects will receive ReDS™ test during hospitalization, at discharge, several home visits and 3 times outpatient follow-up.
  For home visits frequency, ReDS™ tests will be performed every 7 days within 1 month of discharge; at the 2nd to 3rd month, ReDS™ test wil be performed every 15 days. Then ReDS™ test will be performed every 30 days from 4th to 12th months.
  Patients will be followed up in outpatient at 3 months, 6 months, and 12 months after discharge.
  Interventions: Device: ReDS-Guided
- Randomized Arm-Control Group (Sham Comparator): Management of subjects based on standard of care(signs, symptoms, weight, biomarkers, etc.) without lung fluid content information.
  All subjects will receive ReDS™ test during hospitalization, at discharge, several home visits and 3 times outpatient follow-up.
  For home visits frequency, ReDS™ tests will be performed every 7 days within 1 month of discharge; at the 2nd to 3rd month, ReDS™ test wil be performed every 15 days. Then ReDS™ test will be performed every 30 days from 4th to 12th months.
  Patients will be followed up in outpatient at 3 months, 6 months, and 12 months after discharge.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: ReDS-Guided — ReDS™ measurements will be shared with the treating clinicians to guide diuretic treatment when discharge, home visit and outpatient follow-up, but blinded to the subjects.
  At discharge:① If the ReDS™ reading <36%, discharge as planned; ②ReDS™ reading ≥36%, increase the oral diuretic dose, discharge as planned.
  When home visit and outpatient follow-up: ① If the ReDS™ reading <20%, hold diuretics; ② If the ReDS™ reading was between 21-35%, maintain current diuretic dose and optimize GDMT. If the ReDS™ change ≥ 6% from the previous one, increase diuretic dose and optimize the GDMT; ③ If the ReDS™ reading was between 36-45%, increase diuretics and optimize the GDMT, then repeat ReDS™ test after 1 week(home visit); ④ If the ReDS™ reading was above 46%, consider intravenous diuretic therapy, and repeat ReDS™ test after 1 week(home visit) or hospitalization.
  Arms: Randomized Arm-Treatment Group
Other: Usual care — ReDS measurements will not be shared with the treating clinicians and the subjects, diuretic treatment will only be guided using standard clinical care.
  Arms: Randomized Arm-Control Group

SUMMARY:
This clinical study is a multicenter, randomized, controlled clinical study to evaluate the effectiveness of using the noninvasive lung fluid monitoring system based on remote dielectric sensing in guiding the treatment of heart failure.

DETAILED DESCRIPTION:
The main purpose of this study is to explore and validate the effectiveness by using ReDS™ to guide the treatment of heart failure patients during hospitalization and after discharge based on current routine treatment.

The study is divided into two stages

1. Stage 1 is the observation stage for selected heart failure patients during the hospitalization period (from enrollment to discharge). During this stage, patients complete screening, enrollment, and randomization within 72 hours after admission, and are randomly assigned to the experimental group or control group in a 1:1 ratio. All patients receive ReDS™ measurement on the day after randomization, but without using measurement data to intervene the treatment during hospitalization. The randomization of patients and the measurement data remained blind to the treatment clinicians.
2. Stage 2 is the intervention stage, which lasts for 12 months. Firstly, two groups of patients receive ReDS™ measurement on the day of planned discharge. For the control group, this measurement data will still not used as a reference for discharge decision, and remains blind to clinicians; For the experimental group, treatment clinicians will give interventional therapy based on the ReDS™ results.

Approximately 1000 patients will be randomly assigned to the experimental group or control group in a 1:1 ratio, with 500 patients in each group.

Primary/secondary endpoint analysis: will be based on all randomized patients (i.e. ITT population). The Kaplan Meier method was used to estimate the median TTF for each study group. Using the Cox regression model, calculate the regression coefficients or HR values, and their 95% CI. Using forest maps (including HR estimates) to evaluate the homogeneity of intervention effects in important subgroups. The predetermined subgroup analysis will provide additional detailed information in SAP. The hypothesis of primary and secondary endpoints will be formally tested using SAS and Stata statistical software at a unilateral significance level of 0.025.

Safety analysis: Randomized safety analysis based on the safety analysis population.

ELIGIBILITY:
Inclusion criteria:

1. 21 to 85 years old;
2. Sign an informed consent form;
3. The patient is able to comply with the research protocol;
4. Hospitalized due to acute heart failure. The diagnosis of acute heart failure must simultaneously meet the following criteria:

1) Difficulty breathing during screening due to rest or activity; 2) Chest X-ray or chest CT shows clinical manifestations such as pulmonary congestion, pulmonary edema, and pleural effusion; 3) After the onset of this disease and before screening, any test meets the following criteria: BNP ≥ 400 pg/mL or NT proBNP ≥ 1600 pg/mL in patients with sinus rhythm, BNP ≥ 600 pg/mL or NT proBNP ≥ 2400 pg/mL in patients with atrial fibrillation; 4) Intravenous diuretic treatment is required.

Exclusion criteria:

1. Respiratory difficulties caused by non cardiac reasons;
2. Evaluate whether the body condition is not suitable for wearing a ReDS™ non-invasive lung water measuring instrument, including but not limited to: BMI<20 or>39kg/m², height<150cm or>195cm, or flail chest (for patients with BMI between 20-22kg/m², or height between 150-155cm, ReDS™ testing is required to ensure that the body condition is suitable);
3. With a history of heart transplantation or left ventricular assist device implantation, and is still in implantation status;
4. Combination of pulmonary diseases, such as active pneumonia, acute pulmonary embolism, or a history of acute pulmonary embolism within the past 6 months;
5. Severe pulmonary hypertension caused by non left heart disease (pulmonary artery systolic pressure measured by echocardiography ≥ 70mmHg);
6. Simple right heart failure;
7. Patients who undergo thoracotomy or other surgeries or procedures during their intended hospitalization or within one year that affect the wearing of ReDS™;
8. Severe renal insufficiency (eGFR<20ml/min/1.73m²) or dialysis patients;
9. Those with malignant tumors or other serious diseases and an expected survival period of less than 1 year;
10. Pregnant women, pregnancy is defined as the state in which a woman becomes pregnant until the termination of pregnancy;
11. Unable to follow the research instructions or follow the examination, evaluation, and follow-up procedures (including inability to conduct regular follow-up or pulmonary fluid measurement due to the distance from residence to the research center);
12. Any other medical situation that the researcher believes may be a risk to the patient or affect the research results, or any medical situation that the researcher believes is not suitable for the study, including drug or alcohol abuse or mental illness that affects the patient's ability to comply with the protocol or follow-up procedures;
13. Participating in other interventional studies (including patients during washout period).

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The number of cardiovascular deaths | 12 months post-discharge.
The number of recurrent heart failure readmissions | 12 months post-discharge.
  A heart failure readmission is defined as a hospitalization due to worsening heart failure or an emergency department visit requiring intravenous diuretic treatment. If a patient in the ReDS-Guided group is suggested to receive intravenous diuretic based on the ReDS™ home visit , it should not be recorded as an event of heart failure (as this is part of the planned follow-up).
The change of KCCQ score | 12 months post-discharge.

SECONDARY OUTCOMES:
Cardiovascular readmissions | 12 months post-discharge.
  The number of recurrent cardiovascular readmissions.
all-cause mortality | 12 months post-discharge.
  The number of all-cause deaths
First time heart failure readmission | 12 months post-discharge.
  The time from discharge to first heart failure readmission.
All-cause readmissions | 12 months post-discharge.
  The number of recurrent all-cause readmissions.
Cardiovascular mortality | 12 months post-discharge.
  The number of cardiovascular deaths.
All-cause mortality | 12 months post-discharge.
  The number of all-cause deaths.
Change of NT-proBNP | 12 months post-discharge.
  The change of NT-proBNP measurements.

OTHER OUTCOMES:
Total medical costs in the short term (during clinical trials) | 12 months post-discharge.
  Health economics evaluation endpoint
Short term (clinical trial period) total QALY | 12 months post-discharge.
  Health economics evaluation endpoint
Incremental Cost Effect Ratio (ICER) | 12 months post-discharge.
  Health economics evaluation endpoint

IPD SHARING:
Plan to Share IPD: No